CLINICAL TRIAL: NCT00226408
Title: Randomized, Multicenter Study for Adjuvant Treatment of Stage III Malignant Melanoma: Intermittent, High-Dose Intravenous Interferon Alpha-2b Versus Standard High-Dose Interferon Alpha-2b Therapy
Brief Title: Standard High-Dose Alpha Interferon Versus Intermittent High-Dose Alpha Interferon
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dermatologic Cooperative Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-ADJ-5
Record Dates: First submitted 2005-09-25; First posted 2005-09-27 (Estimated); Last update posted 2006-06-21 (Estimated); Status verified 2005-09

CONDITIONS: Adjuvant; Stage III Malignant Melanoma; Interferon Alpha; Therapy
Keywords: melanoma,adjuvant therapy,stageIII Interferon; high dose
MeSH Terms: conditions — Melanoma | interventions — Introns

INTERVENTIONS:
Drug: Interferon-alpha-2b

SUMMARY:
The study protocol is being conducted to compare intermittent high-dose i.v. administation of interferon alpha-2b with the standard high-dose treatment by Kirkwood with distant metastasis free survival (DMFI) as a primary endpoint.

DETAILED DESCRIPTION:
Arm A: Interferon-alpha-2b 20 MIU/m2 for 4 weeks. 5 days a week i.v followed by 48 weeks of treatment with 3 x 10 MIU/m2 s.c Arm B: Interferon-alpha-2b 20 MIU/m2 for 4 weeks. 5 days a week i.v repeated 3 times with 12 treatment-free-weeks between the cycles

Secondary endpoints: Improved overall survival rate, Assess side effects of therapy in both treatment arms, Assess time spent on sick leave, Assess number of treatment-related days in hospital, Assess overall performance status, Assess blood MX protein levels

ELIGIBILITY:
Inclusion Criteria:

* Histological documentet cutaneous malognant melanoma
* Stage IIIa, IIIb, IIIc (AJCC 2002)
* R0 resection dating back no longer than 56 days
* Performance status (ECOG o-1)
* Bone marrow funktion: White cell count > 3000 cells/ul, platletts > 100000 cells/ul, hemoglobin > 10 g/dl
* Liver and kidney funktion: Serum creatinin < 1.5 times upper limit of normal, AST and ALT < 2.5 times upper limit of normal, Serum bilirubin < 2 times upper limit of normal
* Written inform consent

Exclusion Criteria:

* Confirmed distant metastasis
* Choroid or mucosal melanoma
* Pregnant or lactating women and women of childbearing potential not using a reliable form of contraception
* Active autoimmun disease
* patients with history of neuropsychiatric disease requiring hospitalization
* Severe medical condition such us:
* Florid hepatitis
* Severe acute infection
* Myocardial infarction within the past year,symptomatic angina pectoris
* Grade III to IV congestive heart failure
* serious pulmonary disease
* HIV-positive patients with an AIDS - defining condition
* treatment in another clinical drug trial within the last 30 days
* A history of hypersensitivity to interferon alfa
* History of maignant disease during the past 5 years (except for curatively treated skin carcinoma or in situ carcinoma)
* Prior high dose interferon alfa therapy.Prior adjuvant low dose or intermediate-dose interferon alfa therapy is allowed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-11; Study Completion 2005-09

PRIMARY OUTCOMES:
distant metastasis free survival/(DMFI )

SECONDARY OUTCOMES:
overall survival
time to progression
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mohr, MD, Principal Investigator — Elbeklinikum, Buxtehude, Germany; Peter von Wussow, MD, Principal Investigator — 30159 Hannover,Georgstr.46
Locations (13):
- Germany (13):
  - Universitätshautklinik ,St.Josef- Hospital, Bochum
  - Elbekliniken Buxtehude, Buxtehude
  - Universitätshautklinik Köln, Cologne
  - Universitätshautklinik Essen, Essen
  - Universitätsklinik Eppendorf, Hamburg
  - Praxis, Hanover
  - Universitätshautklinik Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Hautklinik, Homburg/ Saar
  - Christian- Albrechts- Universität ,Hautklinik, Kiel
  - Universitätshautklinik Mainz, Mainz
  - universitätsklinikum Münster, Münster
  - Städtische Kliniken Oldenburg, Oldenburg
  - Universitätshautklinik Ulm, Ulm

REFERENCES:
- [Derived] Mohr P, Hauschild A, Trefzer U, Enk A, Tilgen W, Loquai C, Gogas H, Haalck T, Koller J, Dummer R, Gutzmer R, Brockmeyer N, Holzle E, Sunderkotter C, Mauch C, Stein A, Schneider LA, Podda M, Goppner D, Schadendorf D, Weichenthal M. Intermittent High-Dose Intravenous Interferon Alfa-2b for Adjuvant Treatment of Stage III Melanoma: Final Analysis of a Randomized Phase III Dermatologic Cooperative Oncology Group Trial. J Clin Oncol. 2015 Dec 1;33(34):4077-84. doi: 10.1200/JCO.2014.59.6932. Epub 2015 Oct 26. PMID 26503196
- See also: Related Info — http://www.ADO-homepage.de